CLINICAL TRIAL: NCT00870974
Title: Evaluation of [18F]PEB and Positron Emission Tomography (PET) as a Marker of mGluR5 in Subjects w/ Neuropsychiatric Conditions
Brief Title: A PET Brain Imaging Study of mGluR5 in Subjects With Neuropsychiatric Conditions
Acronym: FPEB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, David Russell, MD, PhD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FPEB
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson Disease; Huntington Disease; Autistic Spectrum Disorders; Fragile X Syndrome; Alzheimer Disease; Mild Cognitive Impairment
Keywords: Parkinson; Huntington's; Fragile X; Autistic Spectrum; Alzheimer's; MCI
MeSH Terms: conditions — Parkinson Disease; Huntington Disease; Autism Spectrum Disorder; Fragile X Syndrome; Alzheimer Disease; Cognitive Dysfunction | interventions — Fluorine-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [18F]FPEB and PET imaging (Experimental): To assess [18F] FPEB and PET imaging in subjects with neuropsychiatric conditions.
  Interventions: Drug: [18F]FPEB

INTERVENTIONS:
Drug: [18F]FPEB — Each subject will receive a bolus injection targeted to be 5 mCi and not to exceed 5.5 mCi (not >10% of 5 mCi limit) of [18F]F-PEB
  Other Names: Fluorine-18

SUMMARY:
Measurement of metabotropic glutamate receptor type 5 (mGluR5) binding capacity in the brain, may be a valuable tool in the early detection, understanding, or evaluation of Parkinson disease (PD), Huntington disease (HD), Fragile X syndrome (FXS), Autism Spectrum Disorder(ASD), Alzheimer's Disease(AD), and subjects with mild cognitive impairment (MCI).

The goal of this study is to assess [18F]F-PEB positron emission tomography (PET) imaging as a tool to detect mGluR5 density in the brain of PD, HD, FXS ASD, AD, and MCI research participants and similarly aged healthy subjects.

DETAILED DESCRIPTION:
Informed consent will be obtained for all subjects. All subjects will undergo a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. All subjects will undergo [18F]F-PEB PET imaging. Subjects may also be asked to undergo standard brain MRI to assist in the analysis of the PET images obtained.

ELIGIBILITY:
Written informed consent must be obtained For all females of child-bearing potential, a negative urine or blood pregnancy test on day of [18F]PEB injection.

INCLUSION CRITERIA:

PD subjects:

* Age 30 years or older.
* Clinical diagnosis of PD with at least two of three of the cardinal symptoms of PD (rest tremor, rigidity, bradykinesia)
* Hoehn and Yahr[35] ≤ 4.

HD subjects:

* Age 18 years or older.
* Participants have a clinical diagnosis of symptomatic HD with genetic confirmation
* Subject is able to provide informed consent as judged by the investigator, or assent can be obtained from the subject and informed consent provided by the appropriate legal representative or next of kin.

Healthy volunteers should be 18 years of age or older and have a negative history of neurological or psychiatric illness.

ASD and/or FRAGILE X:

* Age 18 years or older
* Clinical diagnosis of ASD and/or FXS
* Diagnosis of FXS based on gene testing or diagnosis of ASD based on DSM-IV criteria

AD subjects:

* Participants have a positive assessment for dementia of Alzheimer type in accordance with the DSM-IV-TR and probable AD according to the NINCDS-ADRDA criteria.
* Participants do not fulfill the ICC criteria for probable DLB, the NINDS-AIREN for probable vascular dementia, or the Neary criteria for FTD.
* CDR score of 0.5, 1 or 2.

MCI subjects:

* Participants must have a complaint of memory loss, objective impairment in at least one cognitive domain, essentially preserved activities of daily living, and do not meet diagnostic criteria for AD or other form of dementia. Participants do not fulfill the ICC criteria for probable DLB, the NINDS-AIREN for probable vascular dementia, or the Neary criteria for FTD.
* CDR score of ≤ 0.5.

AD and MCI:

* Age 50 years or older.
* MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease. Exclusion criterion may be waived if, in the judgment of the investigator (1) vascular dementia is clinically unlikely and (2) the subject is deemed unable to tolerate the MRI procedure due to claustrophobia, etc.

EXCLUSION CRITERIA:

PD, HD and ASD and/or Fragile X subjects:

* Clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* Any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Clinically significant evidence of vascular disease or alternative neurologic disorder

Healthy volunteers:

* Clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* Any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.

AD and MCI subjects:

* The subject has clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including significant gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Does FPEB reliably represent the known distribution of MGLUR5 in the brain? | at completion of scans

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States